CLINICAL TRIAL: NCT01345838
Title: Acetabular Labral Tear in Dysplastic Hips
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: PAO and labrum
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Developmental Dysplasia of the Hip; Labrum
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dysplasia: Patients with developmental dysplasia of the hip undergoing PAO
  Interventions: Procedure: labrum

INTERVENTIONS:
Procedure: labrum — Two years follow-up after PAO, to find any differences among patients with and without known acetabular labral tears

SUMMARY:
A prospective case-control study of the clinical and radiographic outcome of periacetabular osteotomy in patients with and without preoperative acetabular labral tears.

ELIGIBILITY:
Inclusion Criteria:

* Developmental dysplasia of the hip

Exclusion Criteria:

* contraindication for magnetic resonance arthrography
* severe deformities of the femural head

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients with developmental dysplasia of hip and who is scheduled for PAO
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Prof. D.Msc, Study Chair — Orthopedic Research Unit, Aarhus University Hospital; Charlotte Hartig-Andreasen, MD, Principal Investigator — Orthopedic Research Unit, Aarhus University Hospital
Locations (1):
- Orthopaedic department, Aarhus Universityhospital, Aarhus, Denmark